CLINICAL TRIAL: NCT00288886
Title: Reinforcement of Abstinence and Attendance in Substance Abuse Treatment
Brief Title: Reinforcement of Abstinence and Continuing Care in Substance Abuse Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIR 03-267
Record Dates: First submitted 2006-02-06; First posted 2006-02-08 (Estimated); Results first posted 2014-10-29 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2014-07

CONDITIONS: Substance Use Disorders; Alcohol Abuse; Alcoholism; Substance Dependence; Substance Abuse
Keywords: Compliance; Aftercare; Reinforcement, social; Alcoholics Anonymous; Support Groups; Treatment Outcome
MeSH Terms: conditions — Substance-Related Disorders; Alcoholism; Patient Compliance | interventions — Contracts

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Contracts, Prompts and Reinforcement arm (Experimental): Participants were provided with contracting, prompting and reinforcement of continuing care attendance and substance use abstinence.
  Interventions: Behavioral: Contracting, Prompting and Reinforcement arm
- Control Arm (Active Comparator): Participants were provided with routine care- they did not receive contracting, prompting and reinforcement of continuing care attendance and substance use abstinence.
  Interventions: Behavioral: Control arm

INTERVENTIONS:
Behavioral: Contracting, Prompting and Reinforcement arm — Contracting, prompting and reinforcement of continuing care and abstinence.
  Arms: Contracts, Prompts and Reinforcement arm
Behavioral: Control arm — Routine residential treatment and orientation to continuing care.
  Arms: Control Arm

SUMMARY:
The Contracts, Prompts, and Social Reinforcement (CPR) intervention was designed to address the continuing care adherence needs of veterans presenting for substance use disorder (SUD) treatment. Final results of our recently completed HSR&D clinical trial suggest CPR meaningfully impacts aftercare adherence and abstinence rates. However, CPR did not impact abstinence rates at earlier follow-up points, other important measures of treatment outcome, or AA/NA support group attendance. Furthermore, the generalizability of CPR to other sites has not been established. Thus, the intervention has been modified and pilot testing of this improved version of CPR, which includes contingent reinforcement of abstinence and improved prompting of AA/NA attendance (CPR+), shows promising results. We are conducting a multi-site randomized clinical trial to examine the effectiveness of CPR+. We recruited 183 veterans seeking residential treatment at the Salem and Jackson VAMCs. Our primary hypothesis is that the CPR group will have higher 1-year abstinence rates compared to the STX group. Our secondary hypotheses are that the CPR will be particularly effective for individuals with co-morbid psychiatric disorders, and that the CPR+ group will remain in AA/NA and in aftercare for a longer duration, have fewer days of substance use, fewer hospitalizations, and lower costs of care. Treatment outcome will be measured 3-, 6-, and 12-months after participants enter treatment and compared to baseline levels. The current study will seek to extend past findings to show longer-term effectiveness of the CPR+ intervention on continuing care adherence and greater impact on treatment outcome. Dissemination and implementation efforts will be ongoing for this brief, inexpensive intervention, which offers an important means to improve participation and outcome for individuals seeking SUD treatment within the VAMC. Data collection and analysis has been completed.

DETAILED DESCRIPTION:
The Contracts, Prompts, and Social Reinforcement (CPR) intervention was designed to address the continuing care adherence needs of veterans presenting for substance use disorder (SUD) treatment. Final results of our recently completed HSR&D clinical trial suggest CPR meaningfully impacts aftercare adherence and abstinence rates. Among CPR participants, 55% met the VA's SUD continuity of care performance measure (attending at least 2 therapy sessions each month for 3 months), compared to 36% of those in standard treatment (STX). On the primary outcome variable, 57% of the participants in the CPR condition were abstinent at the 1-year follow-up compared to 37% of those in STX. Post hoc moderator analyses also indicate that the intervention was particularly effective for participants with co-morbid psychiatric disorders. However, CPR did not impact abstinence rates at earlier follow-up points, other important measures of treatment outcome, or AA/NA support group attendance. Furthermore, the generalizability of CPR to other sites has not been established. Thus, the intervention has been modified and pilot testing of this improved version of CPR, which includes contingent reinforcement of abstinence and improved prompting of AA/NA attendance (CPR+), shows promising results. We conducted a multi-site randomized clinical trial to examine the effectiveness of CPR+ with 2 specific goals: 1) to compare CPR+ to STX on adherence to continuing care (i.e., AA/NA participation and aftercare therapy) and 2) to assess its effect on treatment outcome. We recruited 183 veterans seeking residential treatment at the Salem and Jackson VAMCs. Our primary hypothesis is that the CPR group will have higher 1-year abstinence rates compared to the STX group. Our secondary hypotheses are that the CPR will be particularly effective for individuals with co-morbid psychiatric disorders, and that the CPR+ group will remain in AA/NA and in aftercare for a longer duration, have fewer days of substance use, fewer hospitalizations, and lower costs of care. Treatment outcome will be measured 3-, 6-, and 12-months after participants enter treatment and compared to baseline levels using the Form-90 Interview, the Addiction Severity Index (ASI), questionnaire responses, and substance use screens. Treatment adherence will be measured using VA databases, medical records, therapist ratings, and questionnaire responses. Abstinence rates will be analyzed using a logistic regression model in which the parameters of interest are estimated using Generalized Estimating Equations. Secondary outcomes will be analyzed using both marginal and linear mixed-effects models as appropriate. The current study sought to extend past findings to show longer-term effectiveness of the CPR+ intervention on continuing care adherence and greater impact on treatment outcome. Dissemination and implementation efforts are ongoing for this brief, inexpensive intervention, which offers an important means to improve participation and outcome for individuals seeking SUD treatment within the VAMC.

ELIGIBILITY:
Inclusion Criteria:

Participants were recruited from consecutive veterans who successful complete the 28-day SARRTP at the Salem VAMC and the 21-day SARRTP at the Jackson VAMC. Participants who are uninterested in aftercare, who have unstable housing or other factors that made aftercare participation difficult, will be included to maximize the generalizability of our results.

Exclusion Criteria:

Individuals who did not live within a 60-minute drive, and those who did not have transportation and a work schedule allowing attendance of aftercare were ineligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2007-03; Primary Completion 2009-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Lash, PhD, Principal Investigator — Salem VA Medical Center, Salem, VA
Locations (2):
- United States (2):
  - G.V. (Sonny) Montgomery VA Medical Center, Jackson, MS, Jackson, Mississippi
  - Salem VA Medical Center, Salem, VA, Salem, Virginia

REFERENCES:
- [Result] Lash SJ, Timko C, Curran GM, McKay JR, Burden JL. Implementation of evidence-based substance use disorder continuing care interventions. Psychol Addict Behav. 2011 Jun;25(2):238-51. doi: 10.1037/a0022608. PMID 21443297
- [Result] Lash SJ, Burden JL, Parker JD, Stephens RS, Budney AJ, Horner RD, Datta S, Jeffreys AS, Grambow SC. Contracting, prompting and reinforcing substance use disorder continuing care. J Subst Abuse Treat. 2013 Apr;44(4):449-56. doi: 10.1016/j.jsat.2012.09.008. Epub 2012 Oct 31. PMID 23122489

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 426 Consecutive Graduates Screened for Eligibility, 243 (57%) of those were excluded. [203 (48%) not within a 60-minute drive of aftercare; 15 (4%) no transportation, or aftercare not available due to work schedule; 24 (6%) did not consent; 1 excluded for unknown reason(s)]
Groups:
- Standard Treatment (STX): Control condition: Routine residential treatment and orientation to continuing care.
  An addiction therapist from the participants' treatment program met with each participant for an individual aftercare orientation session during the final 4 days of the initial treatment program and again during the ninth week of aftercare. Individuals were also encouraged to get an AA or NA sponsor during this session.
- Contracts, Prompts and Reinforcement (CPR): Contracting, Prompting & Reinforcing Abstinence & Attendance: Contingent reinforcement of abstinence and prompting of AA/NA attendance
  CPR participants received the STX aftercare orientation except they were also provided with the contracting intervention during the orientation sessions, as well as the prompting and reinforcement components of the intervention.
  * Contracting. Participant's completed a behavioral contract for continuing care participation that took approximately 20 minutes to complete during their final 4 days in initial treatment and after 9 weeks of participation in continuing care.
  * Prompting. CPR participants received prompts (mailed appointment cards, telephone reminders) to attend all of their aftercare appointments and AA/NA meetings, and following missed aftercare sessions for 1 year (or until discharged from treatment).
  * Reinforcement. CPR participants received social reinforcement (certificates, honor roll) for attending group therapy.
Period: Overall Study
Arm/Group | Standard Treatment (STX) | Contracts, Prompts and Reinforcement (CPR)
Started | 91 | 92
3-month Follow Up | 82 | 85
6-month Follow Up | 85 | 84
12-month Follow Up | 80 | 81
Completed | 80 | 81
Not Completed | 11 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Treatment (STX) | Contracts, Prompts and Reinforcement (CPR) | Total
Number analyzed (Participants) | 91 | 92 | 183
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.63 (7.88) | 49.55 (8.63) | 50.09 (8.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 88 | 87 | 175
Region of Enrollment [Number; unit: participants]
  United States | 91 | 92 | 183

OUTCOME MEASURES:

1. Primary Outcome: Abstinence Rate (During the Preceding 90 Days) at 12 Months Follow-up Point as Assessed by the Form-90
Description: Participants who were abstinent was assessed via Form-90 Interview (Form 90I) is a structured interview that assesses substance use and related behaviors over the previous 90 days employing a calendar-based follow-back method that provides continuous measures of substance use, and has good reliability. Measures include days abstinent, days using alcohol, days using drugs, total number of standard drinks, and days of self help meeting attendance. Briefer versions were constructed to collect data via telephone in instances when participants did not return for in-person interviews. As a reliability check on participants' self-report, a collateral interview was employed when contacting informants. Participants who denied use on the Form-90, but had a positive substance use screen were considered to be not abstinent for that follow-up point.
Time Frame: Assessed at 12 months
Measure: Number; unit: participants
Arm/Group | Standard Treatment (STX) | Contracts, Prompts and Reinforcement (CPR)
Number analyzed (Participants) | 83 | 81
participants
  Abstinence from alcohol and drugs | 40 | 38
  Abstinence from alcohol | 47 | 51
  Abstinence from drugs | 55 | 49

2. Secondary Outcome: Abstinence Rate (During the Preceding 90 Days) at 3- and 6-months Follow-up Point as Assessed by the Form-90
Description: as for outcome 1
Time Frame: Assessed at 3 and 6 months
Measure: Number; unit: participants
Arm/Group | Standard Treatment (STX) | Contracts, Prompts and Reinforcement (CPR)
Number analyzed (Participants) | 91 | 92
participants
  Abstinence from alcohol and drugs (3 month) | 57 | 57
  Abstinence from alcohol (3 month) | 65 | 69
  Abstinence from drugs (3 month) | 64 | 62
  Abstinence from alcohol and drugs (6 months) | 43 | 43
  Abstinence from alcohol (6 month) | 50 | 61
  Abstinence from drugs (6 month) | 51 | 55

3. Secondary Outcome: Days Until First Use of Alcohol or Drugs
Time Frame: Baseline to 12 months
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Standard Treatment (STX) | Contracts, Prompts and Reinforcement (CPR)
Number analyzed (Participants) | 91 | 92
days | 200.74 (136.31) | 202.43 (140.46)

4. Secondary Outcome: Aftercare Attendance
Description: Measures of aftercare attendance include: Percentage of participants who attended at least 1 aftercare session; percentage of participants who attended at least 2 aftercare sessions/month for at least 3, 6, 9 and 12 months; and percentage of participants who passed the VAMC's SUD continuity of care performance measure (a benchmark for retention of clients in aftercare for at least two visits each month for 3 months following initial treatment)
Time Frame: Assessed at 3-, 6-, 9-, and 12-months
Measure: Number; unit: percentage of participants
Arm/Group | Standard Treatment (STX) | Contracts, Prompts and Reinforcement (CPR)
Number analyzed (Participants) | 91 | 92
percentage of participants
  Attended at least 1 aftercare session | 97 | 97
  Passed the SUD continuity of care measure | 58 | 70
  Attended at least 3 months of treatment | 64 | 76
  Attended at least 6 months of treatment | 35 | 48
  Attended at least 9 months of treatment | 22 | 35
  Attended at least 12 months of treatment | 10 | 16

5. Secondary Outcome: Self-help Support Group Attendance
Time Frame: Assessed over the past 90 days at 3, 6 and 12 months, and cumulative over 1 year
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Standard Treatment (STX) | Contracts, Prompts and Reinforcement (CPR)
Number analyzed (Participants) | 91 | 92
days
  Days of AA or NA attendance (3 months) | 20.18 (21.16) | 23.44 (22.29)
  Days of AA or NA attendance (6 months) | 18.14 (25.90) | 21.99 (26.50)
  Days of AA or NA attendance (12 months) | 12.41 (21.57) | 14.18 (23.21)
  Total Days of AA or NA attendance at 1 year | 45.7 (57.3) | 54.6 (58.2)

6. Secondary Outcome: Days of Substance Abuse (Across the Prior 90 Days)
Time Frame: Assessed at Baseline, 3-, 6-, and 12-month follow-up
Measure: Mean (Standard Deviation); unit: percentage of 90 days
Arm/Group | Standard Treatment (STX) | Contracts, Prompts and Reinforcement (CPR)
Number analyzed (Participants) | 91 | 92
percentage of 90 days
  % of days using alcohol or drugs (Baseline) | 51 (33) | 58 (29)
  % of days using alcohol or drugs (3 month) | 6 (17) | 7 (19)
  % of days using alcohol or drugs (6 month) | 11 (23) | 8 (19)
  % of days using alcohol or drugs (12 month) | 15 (28) | 15 (31)

7. Secondary Outcome: Rates of Hospitalization (Across the Prior 90 Days)
Description: Number of days hospitalized for any reason per the previous 90 days
Time Frame: Assessed at Baseline, 3-, 6-, and 12-months
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Standard Treatment (STX) | Contracts, Prompts and Reinforcement (CPR)
Number analyzed (Participants) | 91 | 92
days
  Days of hospitalization (Baseline) | 9.23 (14.42) | 6.87 (12.39)
  Days of hospitalization (3 months) | 1.18 (4.74) | 1.93 (8.21)
  Days of hospitalization (6 months) | 2.14 (8.74) | 4.23 (14.73)
  Days of hospitalization (12 months) | 1.47 (4.07) | 2.08 (11.27)

ADVERSE EVENTS:
Time Frame: 1 year.
Description: No Adverse Events were found in this behavioral intervention study.
Arm/Group | Standard Treatment (STX) | Contracts, Prompts and Reinforcement (CPR)
Serious Adverse Events (participants affected / at risk) | 0/91 | 0/92
Other Adverse Events (participants affected / at risk) | 0/91 | 0/92

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes